CLINICAL TRIAL: NCT05820282
Title: Using IF-THEN Plans to Increase Healthcare Professional Delivery of Behaviour Change Interventions During Routine Healthcare
Brief Title: Using IF-THEN Plans to Increase Behaviour Change Intervention Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Chris Keyworth, Lecturer in Psychology, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PSYC-398
Record Dates: First submitted 2023-03-22; First posted 2023-04-19 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants in the control condition are presented with a table with two columns containing the same situations and solutions that participants in the experimental group see. Each situation and solution has a radio button (i.e. a tick box) next to it; participants in the control condition are asked to identify situations and solutions and place a tick next to each one they think would be useful to them. Therefore, participants in the control condition are not asked to form implementation intentions.
  Interventions: Other: Control condition
- Intervention (volitional help sheet) (Experimental): Participants in the experimental condition are presented with a table with two columns and nine rows. Nine situations (barriers to delivering behaviour change interventions) are presented in the left hand column and nine solutions (or appropriate responses; processes of change) are presented in the right hand column (as separate drop down menus). Participants in this condition are asked to form implementation intentions by linking critical situations with appropriate responses by choosing an appropriate response from the drop down menu for each critical situation. Participants are told they can make as many situation-solution links as they wanted.
  Interventions: Behavioral: Volitional help sheet

INTERVENTIONS:
Behavioral: Volitional help sheet — Participants are asked to choose from a list of strategies for increasing delivery of behaviour change interventions
  Arms: Intervention (volitional help sheet)
Other: Control condition — Participants are asked to identify situations and solutions and place a tick next to each one they think would be useful to them. Therefore, participants in the control condition are not asked to form implementation intentions.
  Arms: Control

SUMMARY:
The aim of the present research is to test the effectiveness of an implementation intention-based intervention for increasing healthcare professional delivery of behaviour change interventions during routine healthcare.

Each participant will be randomly allocated to one of two conditions. The two conditions are: (1) a control condition, and (2) intervention (form multiple implementation intentions from a drop-down menu). The main outcome measure will be use of face coverings.

DETAILED DESCRIPTION:
Background and study aims

Public health policies are used to compel healthcare professionals to deliver health behaviour change interventions during routine practice. Making Every Contact Count, a National Health Service (NHS) policy aimed at patient-facing healthcare professionals, places prevention at the centre of every NHS patient-HCP contact. Our previous research showed decreasing levels of healthcare professional delivery of health behaviour change interventions. The investigators were also able to provide recommendations for interventions to support healthcare professionals' capabilities, opportunities and motivations in order to sustain delivery of behaviour change interventions in the long term. One key recommendation was that interventions designed to bolster people's "automatic motivation" (i.e., habits, emotions) would likely lead to increased delivery of behaviour change interventions.

Our recent qualitative research suggests enhancing healthcare professionals' capabilities to deliver behaviour change interventions could focus on providing the necessary support to capitalize on the opportunities created by new technology-based approaches to healthcare consultations in light of COVID-19. One such approach may be to support healthcare professionals in identifying patients' barriers to behaviour change, and linking them with possible enablers.

Automatic motivation may be a key intervention target, yet more research is needed to examine effective interventions targeting this. There is a long track record of research showing that implementation intentions are an effective means of changing behaviour, and that such changes in behaviour can be sustained over years. Implementation intentions help people overcome automatic motivation by making the critical situations that may elicit unwanted habits more salient, and ensuring that alternative strategies are deployed. They are best thought of as "if-then" plans: specifying an "if" ensures that triggers to unwanted habits receive greater attention and linking "ifs" with "thens" (e.g., signposting to appropriate information) ensures that the appropriate responses are automatized and replace the unwanted habit. Forming "if-then" plans thus overcome habits.

Aims

To test the effectiveness of an implementation intention-based intervention for increase healthcare professional delivery of behaviour change interventions during routine healthcare.

Who can participate?

Participants were identified from a pre-existing sample of healthcare professionals recruited and incentivised by YouGov (a survey panel company) to complete the questionnaire. The sample was intended to be representative of the patient-facing NHS healthcare professional workforce.

What does the study involve?

Participants complete a series of questionnaires about their experiences delivering health behaviour change interventions during routine healthcare, and are then randomly allocated to one of the two groups. Participants in both conditions are presented with a "volitional help sheet" at the end of the questionnaire. The volitional help sheet was based on previous studies that supported implementation intention formation to support health behaviour change. The specific content of the volitional help sheet (i.e. the barriers and enablers to delivering behaviour change interventions) was based on a qualitative study carried out prior to the present study [ref] and the wider literature [refs]. The volitional help sheet consisted of nine critical situations and nine appropriate responses (labelled "solutions"). The barriers to delivering behaviour change items (i.e. "situations") were translated into "if" statements, for example: "If I believe I don't have a good enough relationship with a patient to talk about healthy lifestyle…"; the processes of change items were translated into "then" statements, for example, "then I would refer to a specialist healthcare professional or another member of my team."

Healthcare professionals in the experimental condition were presented with a table with two columns and nine rows. Nine situations (barriers to delivering behaviour change interventions) are presented in the left hand column and nine solutions (or appropriate responses; processes of change) are presented in the right hand column (as separate drop down menus). Participants in this condition are asked to form implementation intentions by linking critical situations with appropriate responses by choosing an appropriate response from the drop down menu for each critical situation. Participants were told they could make as many situation-solution links as they wanted.

Participants in the control condition were presented with a table with two columns containing the same situations and solutions that participants in the experimental group saw. Each situation and solution had a radio button (i.e. a tick box) next to it; participants in the control condition were asked to identify situations and solutions and place a tick next to each one they thought would be useful to them. Therefore, participants in the control condition were not asked to form implementation intentions.

What are the possible benefits and risks of participating?

By taking part, participants will be helping to understand more about brief interventions to support increased delivery of health behaviour change interventions during routine healthcare. By constructing their own "IF-THEN" plans participants are encouraged to construct their own action plans to deal with potential situations where health behaviour change interventions would be beneficial for their patients.

Below are the main ethical issues and how they will be addressed:

Before giving consent (which will be online, as this is an online-based questionnaire), all project participants will be informed that YouGov will ensure that all data collected is stored confidentially in accordance with their privacy policy.

Participants are still free to withdraw themselves/their data until the data is anonymised (one week after the final follow-up questionnaire). There will be no personally identifiable data in the research publication or in the SPSS file that YouGov send to the research team.

Data will not be shared with any researcher or organisation other than in ways detailed on the PIS. Data (which will be anonymised with no identifiable personal information) may be used for secondary analysis within the research team only.

Who is funding the study?

This study was funded by a research grant obtained through the Research England Policy Support Fund.

Study hypothesis

Current study hypothesis as of 17/03/2023:

The condition that completes a volitional help sheet will report higher delivery of health behaviour change interventions at follow-up than the control condition

Patient information sheet

Not available in web format, please use contact details to request a participant information sheet.

Intervention

Participants complete a series of questionnaires about their experiences delivering health behaviour change interventions during routine healthcare and are then randomly assigned to one of the two conditions:

Participants in the experimental condition are presented with a table with two columns and nine rows. Nine situations (barriers to delivering behaviour change interventions) are presented in the left hand column and nine solutions (or appropriate responses; processes of change) are presented in the right hand column (as separate drop down menus). Participants in this condition are asked to form implementation intentions by linking critical situations with appropriate responses by choosing an appropriate response from the drop down menu for each critical situation. Participants are told they can make as many situation-solution links as they wanted.

Participants in the control condition are presented with a table with two columns containing the same situations and solutions that participants in the experimental group see. Each situation and solution has a radio button (i.e. a tick box) next to it; participants in the control condition are asked to identify situations and solutions and place a tick next to each one they think would be useful to them. Therefore, participants in the control condition are not asked to form implementation intentions.

At each time point participants are asked to report whether they have delivered a health behaviour change intervention to patients to see if the intervention has increased delivery of interventions.

Intervention type

Behavioural

Data analysis plan

Randomisation checks

The investigators will run tests on all outcome and demographic variables to determine if there are any baseline differences in any of these between conditions: chi square will be used for categorical variables and MANOVA for continuous variables.

Mixed ANCOVA (intervention condition (2) x time (3) with baseline behaviour plus confounding factors such as age, gender and healthcare professional group as the covariates) will be used to examine associations between experimental condition (experimental versus control group) and reported delivery of behaviour change interventions at each time point. Similar analyses will be performed on secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 and over, good verbal and written understanding of English A healthcare professional working in the United Kingdom's NHS

Exclusion Criteria:

Aged under 18 years of age, poor verbal and written understanding of English Not a healthcare professional working in the United Kingdom's NHS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1008 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Delivery of health behaviour change interventions | Change from baseline delivery of health behaviour change interventions at 13 months
  Participants will be asked to rate the extent to which they delivered behaviour change interventions during routine consultations on 0-100% scale using the item, "Of the service users you see in a typical working week, who you think would benefit, with what proportion do you Make Every Contact Count?"

SECONDARY OUTCOMES:
Capability, opportunity and motivation (based on Capability, Opportunity, Motivation-Behaviour model) | Change from baseline Capability, opportunity and motivation at 13 months
  Measured using the Capability, Opportunity, Motivation questionnaire. Each of the items (physical opportunity and social opportunity measured on a 0-100 scale, and automatic motivation, reflective motivation, physical capability, and psychological capability measured on a 0-10 scale) will be analysed separately as these each measure a separate construct. Higher scores indicate higher agreement with statements.
  Measured using the Capability, Opportunity, Motivation questionnaire. Each of the items (physical opportunity and social opportunity measured on a 0-100 scale, and automatic motivation, reflective motivation, physical capability, and psychological capability measured on a 0-10 scale) will be analysed separately as these each measure a separate construct. Higher scores indicate higher agreement with statements.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Leeds, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Reasonable requests for data will be available from the study team on request

REFERENCES:
- [Background] Vogt KS, Johnson J, Conner M, Armitage CJ, Keyworth C. Barriers and enablers to delivering opportunistic behaviour change interventions during the COVID-19 pandemic: A qualitative study in healthcare professionals. Br J Health Psychol. 2023 Sep;28(3):773-792. doi: 10.1111/bjhp.12653. Epub 2023 Feb 23. PMID 36822594
- [Background] Armitage CJ. Evidence that implementation intentions can overcome the effects of smoking habits. Health Psychol. 2016 Sep;35(9):935-43. doi: 10.1037/hea0000344. Epub 2016 Apr 7. PMID 27054302
- See also: Intervention page — https://implementationintentions.com/